CLINICAL TRIAL: NCT05647213
Title: Safety and Feasibility of Autologous Induced Pluripotent Stem Cells of Cardiac Lineage in Subjects With Congenital Heart Disease
Brief Title: Autologous Induced Pluripotent Stem Cells of Cardiac Lineage for Congenital Heart Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HeartWorks, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iPSC-CL-001
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Univentricular Heart; Congenital Heart Disease; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: univentricular; heart disease; iPSC; induced pluripotent stem cell
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated (Experimental): Subjects in Treated arm will receive one dose of Investigational Product. Within this arm are three dose levels. Dose level selection will be determined by product availability subjects have available product and when they can be treated. Dose levels will escalate in order of treatment date.
  Interventions: Biological: iPSC-CL
- Control (No Intervention): Subjects who enroll but do not receive Investigational Product will be placed in the control arm.

INTERVENTIONS:
Biological: iPSC-CL — Autologous IPSCL
  Arms: Treated

SUMMARY:
The goal of this clinical trial is to test the safety of lab-grown heart cells made from stem cells in subjects with congenital heart disease. The main questions it aims to answer are:

* Is this product safe to deliver to humans
* Is the conduct of this trial feasible

Participants will be asked to:

* Agree to testing and monitoring before and after product administration
* Receive investigational product
* Agree to lifelong follow-up Researchers will compare subjects from the same pool to see if there is a difference between treated and untreated subjects.

ELIGIBILITY:
Individuals may be considered eligible for enrollment for Part I of this study (Skin Punch Biopsy) if in the best judgment of the Principal Investigator they will meet eligibility criteria outlined below at the time it is determined acceptable investigational product is available for administration (approximately 9 months post skin punch biopsy). Inclusion and exclusion criteria apply to both the treatment and control arms of the study unless otherwise specified.

Inclusion Criteria

Individuals who meet all the following criteria are eligible for enrollment as study participants:

* Age 18 to 40 years old
* Subject must be able to understand and provide informed consent.
* Univentricular congenital heart disease.
* End-stage systolic heart failure, defined as Class IV according to New York Heart Association (NYHA) with abnormal visually estimated ejection fraction below 40%.
* Prognosis of 1 to 1.5 years survival at time of skin biopsy.
* The patient falls into one of the following categories:

  * Currently listed for heart transplantation at an accredited program in the US but has an expected waiting time for a suitable organ that is likely longer than anticipated life-expectancy.
  * Has been denied access to a heart transplantation at an accredited US institution.
  * Is currently on or planning to be on mechanical support as destination therapy.
* All guideline directed therapy available to the subject has been maximized, for a minimum of 3 months prior to enrollment.
* Adequate social support system that facilitates subject participation in all study required tests and procedures and supports the subject's ability to comply with long-term study requirements.

Exclusion Criteria

Individuals who meet any of the following criteria are not eligible for enrollment as study participants:

* No available autologous iPSC-CL as defined by the manufacturer's release criteria. (This applies to Part II of the study and applies to the treatment arm only.)
* History of symptomatic episodes of cardiac arrythmia requiring cardiac defibrillation or escalation of medications.
* Heart failure with preserved ejection fraction.
* Heart failure due to co-morbid conditions (e.g., amyloidosis, valvular heart disease, refractory anemia).
* QTc greater than 500 ms.
* Stage III or higher chronic kidney disease.
* History of liver cirrhosis.
* History of coronary artery disease.
* Uncontrolled diabetes mellitus.
* Any history of cancer.
* Contraindication for use of amiodarone for up to 3 months (treatment arm only).
* Contraindication for insertion of Insertable Cardiac Monitor.
* Contraindication for placement of LifeVest cardioverter defibrillator.
* Positive serology testing for HIV, Hepatitis B, Hepatitis C or Syphilis.
* Obesity with BMI greater than 30.
* Current alcohol or drug abuse precluding heart transplantation.
* Active infection requiring ongoing treatment.
* Contraindication to anesthesia.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality of the data obtained from the study.
* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* History of non-compliance.
* Inability to be accompanied around the clock for any part of the first 3 weeks post product administration.
* Uncontrolled depression.
* Denied heart transplant due to social determinants.
* Current participation in another cardiac interventional clinical trial that could confound the results of this study.
* Previous heart transplant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Short term safety | 3 months
  The primary safety endpoint is short term safety defined as the rate of new or worsening serious adverse events (SAE) from any System Organ Class (SOC) within 3 months of the iPSC-CL delivery as compared to the control arm.
Feasibility | 12 months
  The primary feasibility endpoint is the percentage of individuals with collected skin cells that meet all iPSC-CL release criteria and the percentage of individuals that have cells delivered.

SECONDARY OUTCOMES:
Long term safety | 2 years
  Long term safety measured as new or worsening serious adverse events for two years after iPSC-CL delivery as compared to the control arm.
Cardiac High Sensitivity Troponin T | 1 month
  Change from baseline in Cardiac High Sensitivity Troponin T at 3 hours (±30 min) and 6 hours (±30 min) after iPSC-CL delivery and at 1 month post-surgery as compared to the control arm.
NT-pro-BNP | 3 months
  Change from baseline in NT-pro-BNP levels at 1 and 3 months post iPSC-CL delivery as compared to the control arm.
Tumor marker levels | Three months from date of treatment and every 12 months after treatment, assessed up to 15 years
  Change from baseline in tumor marker levels (PSA (males only), CA 125, CEA, CA 19-9, alpha-fetoprotein (AFP), CA 195, Alpha Subunit HCG) 3 months and annually after iPSC-CL delivery as compared to the control arm.
Panel Reactive Antibody (PRA) levels | 12 months
  Change from baseline in Panel Reactive Antibody (PRA) levels at 3 and 12 months post-iPSC-CL delivery as compared to the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Nelson, M.D., Ph.D., Study Director — HeartWorks, Inc.
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No